CLINICAL TRIAL: NCT04436042
Title: MyHand 2: An Active Hand Orthosis for Stroke Patients
Acronym: MyHand 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Joel Stein, MD, Professor and Chair of the Department of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAS8104; R01NS115652 (NIH)
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Hemiparesis
Keywords: Stroke; Rehabilitation; Hemiparesis; Robotics
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MyHand Treatment (Experimental): Participants will use the MyHand device during repetitive grasp and release tasks.
  Interventions: Device: MyHand Device

INTERVENTIONS:
Device: MyHand Device — These subjects may be asked to attend 1-40 sessions (approximately 90 mins) to trial a variety of device controls and/or components.

SUMMARY:
This study is designed to further develop and test the hardware and software components of the MyHand device based on user feedback and results from our pilot study. The goal is to refine the device so that is more effective and easier for stroke patients to use to increase their hand function.

DETAILED DESCRIPTION:
From previous experimentation with the MyHand device, the investigators have determined that the device can improve the grasping ability of stroke patients. The investigators now aim to make the controls more intuitive and accurate for the users, to enable subjects to grasp a wider array of objects, to make the donning and doffing of the device easier, and to continue to assess the MyHand as it helps subjects in functional tasks.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* History of stroke(s) with most recent stroke at least six months ago
* Upper extremity weakness with impaired ability to complete daily activities with affected hand
* Full passive range of motion in all digits
* Intact cognition to follow directions
* Gross control of proximal upper extremity musculature

Exclusion Criteria:

* Other neurological conditions besides stroke
* Other orthopedic conditions to affected upper extremity
* Significant spasticity in affected upper extremity that impairs device fit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Device Usability and Utility Questionnaire Score | Up to 1 year at study completion
  Subjects will provide feedback about their perceptions of the device's usability and utility for post-stroke upper extremity recovery. Four questions will be rated on a 5-point Likert scale (1) strongly agree to (5) strongly disagree. Five questions will be rated on a 5-point reverse Likert scale (1) strongly disagree to (5) strongly agree.
  The 9 question survey has a score range of 9-45 with higher scores indicating higher levels of device usability and utility.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stein, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No